CLINICAL TRIAL: NCT02802150
Title: The Effect of Oral Zanthoxylum Schinifolium Seed Oil in Individuals With Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, M.D., Ph.D., Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CTCF2_2014_SC
Record Dates: First submitted 2016-02-17; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Dry Eye Syndromes
Keywords: Zanthoxylum schinifolium seed Oil; soy bean oil; omega-3 fatty acid; dry eye disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zanthoxylum schinifolium seed Oil (Active Comparator): Zanthoxylum schinifolium seed Oil 100% (4g/day)
  Interventions: Dietary Supplement: Zanthoxylum Schinifolium Seed Oil(4g/day)
- soy bean oil (Placebo Comparator): soy bean oil 99.9%, edible dyes 0.01% (4g/day)
  Interventions: Dietary Supplement: Soy Bean Oil;placebo(4g/day)

INTERVENTIONS:
Dietary Supplement: Zanthoxylum Schinifolium Seed Oil(4g/day) — parallel design
  Arms: Zanthoxylum schinifolium seed Oil
Dietary Supplement: Soy Bean Oil;placebo(4g/day) — parallel design
  Arms: soy bean oil

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and safety of 10-weeks oral consumption of Zanthoxylum schinifolium seed Oil (ZSO) in patients with mild dry eye disease.

DETAILED DESCRIPTION:
In this double-blind, randomized and placebo-controlled trial, twenty participants experiencing dry eyes symptoms were recruited, and randomly assigned to consume 4 g/day of either ZSO or soy bean oil (SBO) as placebo for 10 weeks. All participants completed the study. Follow-ups of dry eye symptoms and objective signs, inflammatory and oxidative stress markers, and blood lipid analysis were performed.

ELIGIBILITY:
Inclusion criteria:

* men and women
* 20 to 70 years with dry eye disease
* low tear break-up time (TBUT) (<10 seconds) or low Schirmer score (with application of local anesthetic) (<10mm for 5 min) or presence of corneal and conjunctival damage at the time of screening.
* blood level of triglyceride higher than 150 mg/dL or HDL-cholesterol less than 40 and 50 mg/dL for men and women, respectively.

Exclusion Criteria:

* under the anti-inflammatory eye drops for dry eye (topical steroid and topical cyclosporin)
* hypolipidemic medication within 3 months of study entry
* history of chronic disease
* any clinical trial using an investigative medicinal product within 2 months before the first dose of the present study
* allergic or hypersensitive to any of the ingredients in the test products.
* women who were pregnant or breast feeding
* a history of alcoholism or drug abuse or medical or psychological conditions

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
change from Schirmer test(mm) | baseline, 5weeks, 10 weeks
  Measures to assess differences baseline and after the 5-week and 10-week intervention period
change from tear break-up time(seconds) | baseline, 5weeks, 10 weeks
  Measures to assess differences baseline and after the 5-week and 10-week
change from corneal staining(0 to 5 grade) | baseline, 5weeks, 10 weeks
  Measures to assess differences baseline and after the 5-week and 10-week
change from ocular surface disease index(0 to 100 score) | baseline, 5weeks, 10 weeks
  Measures to assess differences baseline and after the 5-weeks and 10-weeks

SECONDARY OUTCOMES:
change from interleukin-13(pg/mL) | baseline, 10 weeks
  Measures to assess differences baseline and after the 10-weeks
change from interferon-gamma(pg/mL) | baseline, 10 weeks
  Measures to assess differences baseline and after the 10-weeks
change from interleukin-1β(pg/mL) | baseline, 10 weeks
  Measures to assess differences baseline and after the 10-weeks
change from interleukin-17(pg/mL) | baseline, 10 weeks
  Measures to assess differences baseline and after the 10-weeks
change from malondialdehyde(nU/L) | baseline, 10 weeks
  Measures to assess differences baseline and after the 10-weeks
change from low-density lipoprotein(pmol/mg) | baseline, 10 weeks
  Measures to assess differences baseline and after the 10-weeks
change from total cholesterol(mg/dL) | baseline, 10 weeks
  Measures to assess differences baseline and after the 10-weeks
change from triglyceride(mg/dL) | baseline, 10 weeks
  Measures to assess differences baseline and after the 10-weeks
change from high-density lipoprotein cholesterol(mg/dL) | baseline, 10 weeks
  Measures to assess differences baseline and after the 10-weeks
change from low-density lipoprotein cholesterol(mg/dL) | baseline, 10 weeks
  Measures to assess differences baseline and after the 10-weeks

OTHER OUTCOMES:
change from fatty acid composition of erythrocyte membrane | baseline, 10 weeks
  Fatty acid composition(%)
  * Palmitic (C16:0)
  * Palmitoleic (C16:1)
  * Stearic (C18:0)
  * Oleic (C18:1)
  * iso-Oleic (C18:1cis)
  * Linoleic (C18:2)
  * Linolenic (C18:3) --> Measures to assess differences baseline and after the 10-week intervention period.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Clinical Trial Center for Functional Foods, Jeonju, Jeollabuk-do

IPD SHARING:
Plan to Share IPD: Undecided